CLINICAL TRIAL: NCT04346030
Title: Comparison of Ultrasound-guided Corticosteroid Injection Versus Corticosteroid Injection and Hydrodissection for Carpal Tunnel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-01-011C
Record Dates: First submitted 2020-04-09; First posted 2020-04-15 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Triamcinolone Acetonide; Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- steroid and hydrodissection (Experimental): ultrasound guided steroid injection using 1ml of 10mg triamcinolone acetonide (Shincort) mixed with 1ml of 2% lidocaine hydrochloride (Xylocaine) and 8cc NS
  Interventions: Drug: Triamcinolone Acetonide; Drug: lidocaine hydrochloride; Drug: normal saline
- steroid only (Active Comparator): ultrasound guided steroid injection using 1ml of 10mg triamcinolone acetonide (Shincort) mixed with 1ml of 2% lidocaine hydrochloride (Xylocaine)
  Interventions: Drug: Triamcinolone Acetonide; Drug: lidocaine hydrochloride

INTERVENTIONS:
Drug: Triamcinolone Acetonide — ultrasound guided steroid injection using 1ml of 10mg triamcinolone acetonide (Shincort) mixed with 1ml of 2% lidocaine hydrochloride (Xylocaine) and 8cc NS
Drug: lidocaine hydrochloride — ultrasound guided steroid injection using 1ml of 10mg triamcinolone acetonide (Shincort) mixed with 1ml of 2% lidocaine hydrochloride (Xylocaine) and 8cc NS
Drug: normal saline — ultrasound guided steroid injection using 1ml of 10mg triamcinolone acetonide (Shincort) mixed with 1ml of 2% lidocaine hydrochloride (Xylocaine) and 8cc NS
  Arms: steroid and hydrodissection

SUMMARY:
The objective of this study is to investigate the effect of ultrasound guided steroid injection versus ultrasound guided steroid hydrodissection to treat patients with CTS.

DETAILED DESCRIPTION:
This study was a prospective, randomized clinical trial. Patients with CTS were randomly treated with sonographically guided corticosteroid injection (group A); sonographically guided hydrodissection and corticosteroid injection (group B).

Boston Carpal tunnel questionnaire, nerve conduction studies and VAS pain score were performed on initial visit and after 6 weeks and 12 weeks .

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of CTS The diagnosis of CTS was confirmed by electrophysiological tests.

Exclusion Criteria:

presence of thenar atrophy any accompanying orthopedic or neurologic disorders that could mimic CTS such as cervical radiculopathy, polyneuropathy, proximal median nerve entrapment, or thoracic outlet syndrome prior steroid injection into the affected carpal tunnel within 6 months or ever received carpal tunnel surgery history of distal radius fracture pregnancy or lactation regular use of systemic NSAIDs ,corticosteroids or diuretics known allergy to corticosteroids and local anesthetics. impaired cognitive function

-

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-04-17 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
change from baseline in the scores on Boston Carpal tunnel Questionnaire (BQ) | 0, 6, 12 weeks.
  The BQ was interviewed-administered to assess the severity of symptoms and functional status

SECONDARY OUTCOMES:
change from baseline in self reported pain intensity | 0, 6, 12 weeks
  patient were asked to indicate the intensity of their average level of pain for the wrist-hand region, using an 11-point scale, ranging from 0 to 10 (worst pain imaginable)
change from baseline in median nerve distal motor latency | 0, 6, 12 weeks
  the CMAPs were obtained via surface electrodes placed on the abductor pollicis brevis muscle. The active recording electrode was placed on the muscle belly, and the reference electrode was placed on the tendon insertion. The median nerve was stimulated 8 cm proximal to the active recording electrode. Distal motor latencies were measured from the onset of stimulus artifact to the onset of the CMAP
Change from Baseline in sensory nerve conduction velocity | 0, 6, 12 weeks
  SNAPs were obtained using an antidromic method and recorded by surface electrodes placed at the proximal and distal interphalangeal joints of the index finger for the median nerve and the same joints of the little finger for the ulnar nerve. The median nerves were stimulated at the wrist at a distance of 14 cm from the wrist to the active electrode. Distal sensory latencies were measured from the onset of the stimulus artifact to the onset of the SNAP. SNCV was calculated dividing the distance of 14 cm by the distal sensory latency.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei veteran general hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No